CLINICAL TRIAL: NCT04225949
Title: Patients Understanding of PROM Graphs: a Randomized Controlled Trial
Brief Title: Patients Understanding of PROM Graphs
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical Reasons (Research Staff)
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 54088
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- line graph (Experimental)
  Interventions: Other: survey 1
- bar graph (Active Comparator)
  Interventions: Other: survey 2

INTERVENTIONS:
Other: survey 1 — survey with one version of depiction
  Arms: line graph
Other: survey 2 — survey with one version of depiction
  Arms: bar graph

SUMMARY:
This study evaluates patients' ability to understand PROM scores when presented in graphs. One half will receive one version of the survey, while the other half will receive a second version of the survey.

ELIGIBILITY:
Inclusion Criteria:

* patient at Stanford Clinics
* orthopaedic condition

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2040-05-15 (Estimated); Primary Completion 2040-08-01 (Estimated); Study Completion 2040-08-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge test | immediately after completing survey
  Knowledge test questionnaire assessing the ability to understand the information the graphs. scored 0-100% correct

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD